CLINICAL TRIAL: NCT04032223
Title: Patient Satisfaction and Retention in Cast Metal Versus 3D Printed Metal Copings in Implant Supported Mandibular Telescopic Overdenture
Brief Title: Patient Satisfaction and Retention in Implant Supported Telescopic Overdenture With Different Copings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Amr Abdelmoez Abosabaa, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO305
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Implant Supported Telescopic Overdenture
Keywords: 3D printed coping , overdenture, Implant , cast metal

STUDY DESIGN:
Intervention Model Description: It is Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed metal copings (Experimental): 3D printed primary and secondary metal copings inderctly from 3D printed resin in mandibular implant supported telescopic overdenture , Single Implants are placed in the interforaminal region bilaterally .
  Interventions: Procedure: Implant placemet in the mandibular canine regions
- Cast metal copings (Active Comparator): Cast metal primary and secondary metal copings in mandibular implant supported telescopic overdenture , Single Implants are placed in the interforaminal region bilaterally .
  Interventions: Procedure: Implant placemet in the mandibular canine regions

INTERVENTIONS:
Procedure: Implant placemet in the mandibular canine regions — Implant placemet in the mandibular canine regions retained by cast metal copings or 3D printed metal copings to deliver Implant Supported telescopic overdenture in the mandible
  Other Names: Metal copings different designs in implant supported telescopic overdenture

SUMMARY:
Implant retained overdentures provided more satisfaction with regard to conventional denture related problems such as esthetics, speech, chewing, fit and retention, function and quality of life. Evaluation of patient satisfaction allows direct quantification of patients' opinions on different aspects of a given treatment.

Studies have indicated that conventional complete denture wearers rehabilitated with mandibular implant supported overdenture experience better retention and stability, improved overall function and satisfaction.

Patient satisfaction is one factor that influences the success of overdenture treatment(Naert, Alsaadi et al. 2004). Previous studies have shown a difference between patients' satisfaction with their dental prostheses and clinicians' assessments of patients' oral condition.(Emami, Heydecke et al. 2009).This indicates that clinical assessments of dentures are not valid predictors of patient satisfaction.

The two primary methods used to fabricate these restorations may be subtractive (milling and grinding) or additive manufacturing (Rapid Prototype, RP or 3D printing), The 3D printing technology has been incorporated into dentistry, but does not include ceramics and is limited to polymers.

3D printing by rapid prototyping has many advantages which are the availability of high production rate where the technician can easily produce over 150 units per hour. Also the quality control of wax copings which results in high precision fit and constant wall thickness. This will result in better stability and retention and consequently patient satisfaction. Finally is the reduced finishing work needed on cast copings. The irregularities in wax coping thickness can be avoided.

DETAILED DESCRIPTION:
Cast metal coping is the comparator. Because of their parallel walled design, telescopic crowns provide horizontal stability, thus stabilizing the prosthesis against lateral dislodging forces. The overdenture's self finding mechanism in telescopic constructions facilitates prosthesis insertion considerably.

Telescopic constructions seem to be easy to care for as they do not possess areas of difficult access for maintenance. This is why this construction also seems to be an effective treatment modality for geriatric patients with serious systemic diseases, which affect the degree of dexterity.

Despite rapid development in overdenture attachments and implant-supported overdentures with cast metal copings remain a viable and usable modality in dental practice. There is limited clinical follow-up data of the complications associated with overdentures and abutment teeth restored with metal copings, including post-procedural and prosthetic problems.

ELIGIBILITY:
Inclusion Criteria:

Patients' age ranging from 45 -65 years old Patients are males or females Completely edentulous maxilla and mandible. Sufficient restorative space ( Not less than 12mm) Co-operative patient that should show motivation to follow up. Sufficient bone to receive Dental implant 3.7mm diameter and 10 mm length in the interforaminal region.

• Exclusion criteria: Patients having any bony undercuts. Patients having any disease affecting muscle coordination as Parkinsonism. Uncontrolled diabetic patients. Patients having limited mouth opening. Patients having bad oral hygiene.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — patients are eligible for implant placment over 18 years
Enrollment: 20 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 3 months
  Patients will be recalled on their scheduled dates to the Prosthodontics department ,Faculty of Dentistry , Cairo University. The patient-based outcomes that will be used in this thesis included the variables measured on the 100-mm VAS (Visual Analogue Scale) and on Category Scales (CAT) that had been previously validated

SECONDARY OUTCOMES:
Retention | 6 months
  small perpendicular metal tubes were placed a few millimetres underneath the canines in the mandibular denture base.
  In this manner the denture could be rigidly and reproducibly connected to the retention-measuring device. Retention measuring device is a device that was developed to apply an increasing, vertical force on the denture The force was administered througha straight metal bar that was fitted withstrain gauges (Measurements Group Inc.,Raleigh, NC, USA). The bar was rigidly connected to the denture.

CONTACTS AND LOCATIONS:
Overall Officials: Yusr O Mady, PHD, Study Chair — Cairo University; Nancy N Elsherbini, PHD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
I will check with my study chair.

REFERENCES:
- [Background] Yunus N, Saub R, Taiyeb Ali TB, Salleh NM, Baig MR. Patient-based and clinical outcomes of implant telescopic attachment-retained mandibular overdentures: a 1-year longitudinal prospective study. Int J Oral Maxillofac Implants. 2014 Sep-Oct;29(5):1149-56. doi: 10.11607/jomi.3328. PMID 25216142